CLINICAL TRIAL: NCT05292170
Title: Influences of Female Sex and Reproductive Hormones on Physiological Aspects of Heat Acclimation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-07Hc
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Heat Stress, Exertional
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Males (Experimental): 10 consecutive day heat acclimation in males
  Interventions: Other: Heat acclimation
- Females + high hormones (Experimental): 10 consecutive day heat acclimation in females with high hormonal dose
  Interventions: Other: Heat acclimation
- Females + low hormones (Experimental): 10 consecutive day heat acclimation in females with low hormonal dose
  Interventions: Other: Heat acclimation

INTERVENTIONS:
Other: Heat acclimation — 10 consecutive days of heat acclimation

SUMMARY:
Women are often understudied in thermal physiology research, leaving recommendations for Soldier safety and performance in hot conditions based largely on data collected in men. Female sex hormones estradiol and progesterone clearly have non-reproductive physiological effects, including influences on thermoregulatory and cardiovascular function. However, mechanisms of differing physiological adaptations to repeated heat exposure (i.e., heat acclimation) as a function of reproductive hormone status have yet to be investigated in a systematic way. Understanding possible sex differences in adaptation or mechanisms for adaptation during heat acclimation is important to ultimately optimize interventions to maximize soldier health and safety during training and deployment in the heat. Our goals in the present study are to evaluate physiological and biophysical responses to a standard heat acclimation protocol in a group of young, healthy men and women. Thirty individuals (n=10 males, n=10 women with a low hormonal status (i.e. early follicular phase), n=10 women with a high hormonal status (i.e. midluteal phase)) will complete 10 consecutive days of exercise (treadmill walking: 3.1 mph/2% grade) in the heat (40°C /40% relative humidity) up to 3hr per day. Changes in core temperature, heart rate, and sex hormones will be assessed to examine differences in thermoregulatory response to heat acclimation.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females, age 18-40 y (17 y for active duty military)

  * Eumenorrheic females (menstrual cycle length between 24-35 days) or females taking oral contraceptives
  * In good health as determined by OMSO (Office of Medical Support and Oversight) General Medical Clearance and willing to report all medications and dietary supplements (i.e. cold medication, Tylenol. Aleve) to the PI and OMSO.
  * Passed his/her most recent Army Combat Fitness Test (ACFT) (military volunteers only) or exercise at least 2 times per week (civilian volunteers)
  * Willing to not exercise, or drink alcoholic beverages for 24 hours before each testing session
  * Willing to not consume caffeine 12 hours prior to any testing sessions
  * Willing to refrain from additional moderate to strenuous physical activity throughout testing period
  * Males and females with BMI <30

Exclusion Criteria:

* • Females who are pregnant or planning to become pregnant during the study

  * Females utilizing implantable contraception (intrauterine device, implantable bar)
  * Tested positive for COVID-19 within the past 30 days.
  * Taking prescription or over the counter medication, other than a contraceptive (unless approved by OMSO and Principal Investigator (PI))
  * Tobacco users, or anyone who has used tobacco within the last four months
  * Physical problems/injuries that would affect walking or running on a treadmill
  * Allergy to skin adhesive
  * Heart, lung, kidney, muscle, endocrine, or nerve disorder(s)
  * History of heat intolerance or orthostatic intolerance
  * Diagnosed and/or treated for fluid/electrolyte imbalance within the last 30 days
  * History of obstructive disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis.
  * Scheduled MRI during testing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis gender males and females
Enrollment: 27 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Core temperature | 10 days
Heart rate | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States